CLINICAL TRIAL: NCT03536975
Title: Pilot Study to Identify the Benefits CAREGIVERSPRO-MMD Platform Use Based on the Information and Communications Technology, Dedicated to the Support and Assistance of Dyads Living With Neurocognitive Diseases Including Persons Living With Mild Cognitive Impairment or Mild to Moderate Dementia and Their Primary Caregivers
Brief Title: Identify the Benefits CAREGIVERSPRO-MMD Platform Use Based on the Information and Communications Technology, Dedicated to the Support and Assistance of Dyads Living With Neurocognitive Diseases and Their Primary Caregivers
Acronym: CAREGIVERSPRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Collaborators: Centre Hospitalier Intercommunal Elbeuf-Louviers-Val de Reuil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016/369/HP
Record Dates: First submitted 2018-01-30; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Cognitive Impairment, Mild; Dementia, Mild
Keywords: Dementia; Mild Dementia; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Intervention group using the "CAREGIVERSPRO-MMD" platform versus control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platform (Other): Group with access to the web platform "CAREGIVERSPRO-MMD"
  Interventions: Other: Platform
- Control (No Intervention): Group without any access to the web platform

INTERVENTIONS:
Other: Platform — The groups will be comprised of one "intervention" group with access to the web platform "CAREGIVERSPRO-MMD" and another "control" group without any access to it
  Arms: Platform

SUMMARY:
Our main goal is to test a web platform accessible by computers, smartphones and tablets, addressed specifically to caregivers and people with mild cognitive deterioration or mild to moderate dementia providing added value services based on social networks, adapted interventions, clinic strategies and gamification to improve the quality of life of caregivers and people living with dementia (dyads) and permitting to leave in the community as long as possible.

To evaluate the platform effectiveness and impact in dementia type disease affected people and caregivers a randomized, controlled, parallel, longitudinal is proposed. The objective will be to assess during 18 months aspects related to health of individuals (general aspect of health, neuropsychological, daily living functionalities, quality of life, treatment adherence, comorbidities ...), social aspects (improving dyad relationship…) and economics (cost-effectiveness of platform utilization), as well as satisfaction degree and usability of platform.

ELIGIBILITY:
Inclusion Criteria:

* For patients People, aged 50 and over, living in the community, who are able to give informed consent.

Diagnosed with mild cognitive impairment (MCI) according to Petersen criteria or mild to moderate dementia diagnosed according on DSM-IV criteria.

Having a Clinical Dementia Rating (CDR) of 0.5 for MCI, 1-2 for mild to moderate dementia Having a Mini-Mental Exam score (MMSE) between 30 and 25 (inclusive) for MCI, and between 24 and 10 (inclusive) for dementia.

Having a primary caregiver, familiar (or not), informal (or not) identified and also included in the study.

Be willing to use Information Technology and Communications (ICT) according to the investigator criteria.

Affiliated to the social security system.

* For caregivers People, aged 18 years and over, with no diagnosis or no evidence of mild cognitive impairment or mild to moderate dementia (according DSM-IV criteria), who are able to give informed consent and with an intention to complete the study.

Primary caregivers, informal (or not), familiar (or not), of person with mild cognitive impairment or mild to moderate dementia People with Internet access and basic knowledge and skills in managing internet and social networks, or keen to learn, according to the investigator criteria Having a Geriatric Depression Scale (GDS-Yesavage - 15 items) score less than 11 at the time of entry into the trial indicating no severe depressive symptoms or for people < 50 years a MADRS < 15 Having no specific conditions (evaluated by the investigator) reducing their physical abilities below the norm for their age that would limit or impair CAREGIVERSPRO-MMD platform use.

Be willing to use Information Technology and Communications (ICT) according to the investigator criteria Affiliated to the social security system

Exclusion Criteria:

* Terminal or severe illness with survival prognosis less than 18 months
* Not speaking nor reading French
* Enrolled in another clinical trial
* For the patients : Having delusions, hallucinations, behavioural disturbances, that may interfere with the use of Information and Communications Technology (ICT) tools ; Under guardianship and/or under curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Burden of primary caregivers | 18 months
  To evaluate the perceived burden of primary caregivers of persons living with mild cognitive impairment or mild to moderate dementia in order to identify a benefit from use of the CAREGIVERSPRO-MMD platform. The perceived burden will be evaluated by using a 29-item scale, Zarit Burden Interview (ZBI).

SECONDARY OUTCOMES:
Quality of life of patients | 6 months
  The 28-item DEMQoL (Dementia Quality of Life Proxy) assesses quality of life of people with mild to moderate dementia. It evaluates five domains: daily activities and locking after health and well-being, cognitive functioning, social relationships and self-concept.
Quality of life of patients | 18 months
  The 28-item DEMQoL (Dementia Quality of Life Proxy) assesses quality of life of people with mild to moderate dementia. It evaluates five domains: daily activities and locking after health and well-being, cognitive functioning, social relationships and self-concept.
Quality of life of patients | 12 months
  The 28-item DEMQoL (Dementia Quality of Life Proxy) assesses quality of life of people with mild to moderate dementia. It evaluates five domains: daily activities and locking after health and well-being, cognitive functioning, social relationships and self-concept.
Quality of life of caregivers | 6 months
  The SF-36v2 - Medical Outcomes Study (MOS) 36-Item Short Form 2nd version will be used for caregivers.
Quality of life of caregivers | 12 months
  The SF-36v2 - Medical Outcomes Study (MOS) 36-Item Short Form 2nd version will be used for caregivers.
Cognitive symptoms of patients | 18 months
  Mini-Mental State Examination will be used to evaluate cognitive symptoms of patients with mild to moderate dementia.
Cognitive symptoms of patients | 6 months
  Mini-Mental State Examination will be used to evaluate cognitive symptoms of patients with mild to moderate dementia.
Cognitive symptoms of patients | 12 months
  Mini-Mental State Examination will be used to evaluate cognitive symptoms of patients with mild to moderate dementia.
Psychological symptoms of caregivers (1) | 6 months
  Geriatric Depression Scale will be used to evaluate depression of older caregivers
Psychological symptoms of caregivers (1) | 12 months
  Geriatric Depression Scale will be used to evaluate depression of older caregivers
Psychological symptoms of caregivers (1) | 18 months
  Geriatric Depression Scale will be used to evaluate depression of older caregivers
Psychological symptoms of caregivers (2) | 6 months
  State Trait Anxiety Inventory will be used to measure trait and state anxiety of caregivers
Psychological symptoms of caregivers (2) | 12 months
  State Trait Anxiety Inventory will be used to measure trait and state anxiety of caregivers
Psychological symptoms of caregivers (2) | 18 months
  State Trait Anxiety Inventory will be used to measure trait and state anxiety of caregivers
Instrumental Activities of Daily Living | 6 months
  The ability to perform tasks necessary to live independently in the community will be assessed using Lawton Instrumental Activities of Daily Living Scale (IADL), (Lawton and Brody 1969)
Instrumental Activities of Daily Living | 12 months
  The ability to perform tasks necessary to live independently in the community will be assessed using Lawton Instrumental Activities of Daily Living Scale (IADL), (Lawton and Brody 1969)
Instrumental Activities of Daily Living | 18 months
  The ability to perform tasks necessary to live independently in the community will be assessed using Lawton Instrumental Activities of Daily Living Scale (IADL), (Lawton and Brody 1969)
Activities of Daily Living | 12 months
  Performance in activity of daily living will be measured using Barthel Index of Activities of Daily Living scale (BADL) (Mahoney and Barthel 1965).
Activities of Daily Living | 18 months
  Performance in activity of daily living will be measured using Barthel Index of Activities of Daily Living scale (BADL) (Mahoney and Barthel 1965).
Activities of Daily Living | 6 months
  Performance in activity of daily living will be measured using Barthel Index of Activities of Daily Living scale (BADL) (Mahoney and Barthel 1965).
Behavioural-psychological symptoms of patients (1) | 6 months
  Behavioural-psychological symptoms will be evaluated using NeuroPsychiatric Inventory (12-item NPI). The score takes into account the frequency and severity of each behavioural symptom.
Behavioural-psychological symptoms of patients (1) | 12 months
  Behavioural-psychological symptoms will be evaluated using NeuroPsychiatric Inventory (12-item NPI). The score takes into account the frequency and severity of each behavioural symptom.
Behavioural-psychological symptoms of patients (1) | 18 months
  Behavioural-psychological symptoms will be evaluated using NeuroPsychiatric Inventory (12-item NPI). The score takes into account the frequency and severity of each behavioural symptom.
Behavioural-psychological symptoms of patients (2) | 18 months
  Geriatric Depression Scale 15 items evaluate depression of older people. A score above 11 is in favour of depression state.
Behavioural-psychological symptoms of patients (2) | 6 months
  Geriatric Depression Scale 15 items evaluate depression of older people. A score above 11 is in favour of depression state.
Behavioural-psychological symptoms of patients (2) | 12 months
  Geriatric Depression Scale 15 items evaluate depression of older people. A score above 11 is in favour of depression state.
Perceived Social Support | 6 months
  Multidimensional Scale of Perceived Social Support (MSPSS) 12 items scale will be used to assess an individual's perception of the social support received from family, friends and significant others. Each item is quoted from 1(totally disagree) to 7 (totally agree).
Perceived Social Support | 12 months
  Multidimensional Scale of Perceived Social Support (MSPSS) 12 items scale will be used to assess an individual's perception of the social support received from family, friends and significant others. Each item is quoted from 1(totally disagree) to 7 (totally agree).
Perceived Social Support | 18 months
  Multidimensional Scale of Perceived Social Support (MSPSS) 12 items scale will be used to assess an individual's perception of the social support received from family, friends and significant others. Each item is quoted from 1(totally disagree) to 7 (totally agree).
Relationships | 6 months
  The Flourishing Scale will be used to measure of the respondent's self-perceived success in important areas such as relationships, self-esteem, purpose and optimism. The scale provides a single psychological well-being score. It is a 8-item scale quoted from 1(totally disagree) to 7 (totally agree).
Relationships | 12 months
  The Flourishing Scale will be used to measure of the respondent's self-perceived success in important areas such as relationships, self-esteem, purpose and optimism. The scale provides a single psychological well-being score. It is a 8-item scale quoted from 1(totally disagree) to 7 (totally agree).
Relationships | 18 months
  The Flourishing Scale will be used to measure of the respondent's self-perceived success in important areas such as relationships, self-esteem, purpose and optimism. The scale provides a single psychological well-being score. It is a 8-item scale quoted from 1(totally disagree) to 7 (totally agree).

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Landrin, MD, Principal Investigator — University Hospital, Rouen
Locations (2):
- France (2):
  - Centre Hospitalier Intercommunal Elbeuf Louviers, Elbeuf
  - Rouen University Hospital, Rouen